CLINICAL TRIAL: NCT00315484
Title: A Randomized, Open-Label Study Of Epoetin Alfa (PROCRIT) Versus Darbepoetin Alfa (ARANESP) To Evaluate Hematologic Response Rate In Anemic Cancer Patients Receiving Chemotherapy
Brief Title: Hematologic Response of Epoetin Alfa (PROCRIT) Versus Darbepoetin Alfa (ARANESP) in Chemotherapy Induced Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004609
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Chemotherapy
Keywords: Anemia; chemotherapy; hemoglobin level; recombinant human erythropoietin; epoetin alfa; darbepoetin alfa
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa; Darbepoetin alfa

INTERVENTIONS:
Drug: Epoetin alfa and Darbepoetin alfa

SUMMARY:
The purpose of this study is to compare hemoglobin (Hgb) response rates between epoetin alfa (PROCRIT; 40,000 Units (U) SC weekly) and darbepoetin alfa (ARANESP; 200 mcg every other week) in anemic cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy related anemia occurs in a majority of cancer patients and can cause impaired treatment outcomes, increased treatment-related complications and altered quality of life. Epoetin alfa administered on a weekly dosing schedule of 40,000 Units subcutaneously ([SC], under the skin) with dose adjustments based on hematologic response produces significant improvement in hemoglobin levels, decreased transfusion frequency and improved quality of life. It is unknown if the recently developed agent, darbepoetin alfa, administered on an every other week fixed dose will produce similar improvements in hematologic and quality of life outcomes. Thus, further randomization studies are warranted utilizing once weekly dosing (QW) of Epoetin alfa compared to once every other week (Q2W) darbepoetin alfa. Patients will receive study medications for up to 16 weeks.Safety & efficacy evaluations will be performed at specified intervals throughout the study.The study hypothesis is that the Week 5 hemoglobin response rate in the Epoetin alfa group is better than that in the Darbepoetin alfa group. The starting dose for study drug is either Epoetin alfa (PROCRIT) 40,000 Units SC QW or Darbepoetin alfa (ARANESP) 200 mcg SC Q2W. Doses may be adjusted depending on the patient's hemoglobin levels up a maximum of 60,000 IU SC QW Epoetin alfa or 300 mcg SC Q2W Darbepoetin alfa.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a solid tumor malignancy
* Baseline hemoglobin value of <11 g/dL
* Scheduled to receive cyclic chemotherapy for a minimum of 12 weeks
* < 2 prior chemotherapy regimens in a metastatic setting
* Adequate hematologic & renal function and platelet count >100,000/mm3
* Estimated life expectancy of > 6 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2

Exclusion Criteria:

* History of stem cell or bone marrow transplant
* Anemia due to factors other than cancer/chemotherapy
* Prior treatment with epoetin alfa or darbepoetin alfa or any investigational forms of erythropoietin within the previous 3 months
* Significant, uncontrolled disease/dysfunction of the pulmonary, cardiovascular, endocrine, neurologic, gastrointestinal, or genitourinary systems not attributable to underlying malignancy or chemotherapy
* Uncontrolled hypertension or recent history (within 6 months) of uncontrolled cardiac arrhythmias, pulmonary embolism, thrombosis
* new onset of seizures
* history of second active malignancy
* Major infection requiring hospitalization and antibiotics within 14 days of randomization
* Transfusion of white blood cells or packed red blood cells within 28 days of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2003-02; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will evaluate the proportion of patients achieving >1 g/dL hemoglobin increase by week 5.

SECONDARY OUTCOMES:
1) time to hemoglobin (Hgb) increase of 1g/dL; 2) proportion of pts achieving a >1 g/dL Hgb increase by Wk 9; 3) proportion of pts achieving a >2g/dL Hgb increase by Wk 9; 4) Hgb values over time; 5) cumulative RBC transfusion Wk 5 to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.

REFERENCES:
- [Result] Waltzman R, Croot C, Justice GR, Fesen MR, Charu V, Williams D. Randomized comparison of epoetin alfa (40,000 U weekly) and darbepoetin alfa (200 microg every 2 weeks) in anemic patients with cancer receiving chemotherapy. Oncologist. 2005 Sep;10(8):642-50. doi: 10.1634/theoncologist.10-8-642. PMID 16177289
- See also: A Randomized, Open-Label Study of Epoetin Alfa (PROCRIT) Versus Darbepoetin Alfa (ARANESP) to Evaluate Hematologic Response Rate in Anemic Cancer Patients Receiving Chemotherapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=925&filename=CR004609_CSR.pdf